CLINICAL TRIAL: NCT03021057
Title: PD-1 Blockade With Pembrolizumab in Relapsed/Refractory Mature T-cell and NK-cell Lymphomas
Brief Title: Pembrolizumab for T/NK-cell lymphomasNK-cell Lymphomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr. Eric W.C. Tse, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HKU-MK-NKT01
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: T-Cell Lymphoma; NK-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pembrolizumab (Experimental): 200mg i.v. once every 3 weeks Number of Cycles: until progression or unacceptable toxicity develops
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — 200mg i.v. once every 3 weeks Number of Cycles: until progression or unacceptable toxicity develops
  Other Names: Keytruda

SUMMARY:
Conventional chemotherapeutic regimens designed for aggressive B-cell lymphomas are generally less effective when applied to mature T-cell or NK-cell lymphomas. The treatment outcome for relapsed or refractory disease is especially poor.

This is a single centre, prospective, non-randomized, open-label, phase II study to evaluate the efficacy of pembrolizumab in patients with relapsed or refractory mature T-cell or NK-cell lymphomas. Patients will receive pembrolizumab 200mg i.v. once every 3 weeks until disease progression or unacceptable toxicity.

A baseline radiological assessment by positron emission tomography / computed tomography (PET/CT) scan is obtained before commencement of treatment. Tumor response and progression are evaluated by physical examination, standard laboratory tests, and PET/CT scan according to standard criteria. Standard response criteria for non-Hodgkin lymphomas are used for assessment . PET/CT scan will be done at week 12, week 24, week 36 and every 18 weeks thereafter.

DETAILED DESCRIPTION:
Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype against PD-1, designed to directly block its interaction with PD-L1 and PD-L2. KeytrudaTM (pembrolizumab) has recently been approved in the United Stated for the treatment of melanoma that is unresectable or metastatic, or has progressed following ipilumumab and, (if BRAF V600 mutation positive), a BRAF inhibitor.

Mature T-cell and nature killer (NK)-cell lymphomas are lymphoid malignancies that are derived from T-cell and NK-cell lineages. They are less prevalent than B-cell lymphomas. Interestingly, there are distinct geographic differences in their distribution and prevalence. Nodal lymphomas including peripheral T-cell lymphoma, not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), anaplastic large cell lymphoma (ALCL) and cutaneous T-cell lymphomas (CTCL) predominate in Western populations, accounting for about 10% of all lymphomas. In Asian countries, however, extranodal NK/T-cell lymphoma, nasal type, is much more prevalent, constituting 10% of all lymphomas; with AITL, ALCL and PTCL-NOS accounting for another 10%. Epstein Barr virus (EBV) infection is found in all cases of extranodal NK/T-cell lymphomas, the majority of AITL, and a significant proportion of PTCL-NOS, implying that it plays an important pathogenetic role.

Conventional chemotherapeutic regimens designed for aggressive B-cell lymphomas are generally less effective when applied to mature T-cell or NK-cell lymphomas. The treatment outcome for relapsed or refractory disease is especially poor. In a recent retrospective analysis, the median overall survival (OS) and progression-free survival (PFS) in patients with disease relapse were found to be only 5.5 and 3.1 months respectively. The efficacy of newly approved agents such as pralatrexate and romidepsin for relapsed or refractory T-cell lymphomas is modest, with an average overall response rate (ORR) of around 20-30% only. Novel therapeutic approaches are therefore needed for this group of patients with dismal prognosis.

PD-1 blockade using anti-PD1 monoclonal antibody has been shown to be highly effective for relapsed/refractory classical Hodgkin lymphoma. Furthermore, clinical response has also been seen in relapsed T-cell lymphomas after treatment with anti-PD-1 antibody in phase I studies. In addition, previous reports have shown that EBV infection may enhance the expression of PD-L1 in tumour cells, and that some EBV-associated lymphomas such as NK/T-cell lymphoma express high level of PD-L1, suggesting that EBV-associated mature T-cell and NK-cell lymphomas may be more susceptible to PD-1 blockade.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) will be considered on a case-by-case basis.
4. Have a performance status of 0 or 1 on the ECOG Performance Scale.
5. Demonstrate adequate organ function , all screening labs should be performed within 10 days of treatment initiation.
6. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
7. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
8. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has undergone prior allogeneic HSCT
4. Has a known history of active TB (Bacillus Tuberculosis)
5. Has hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B virus or Hepatitis C virus infection.
19. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate (CR) | 12 weeks
  Complete remission (CR) rate at 12 weeks and thereafter

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 weeks
  defined as the proportion of patients achieving CR or PR at 12 weeks and thereafter.
Duration of response (DOR) | 2 years
  defined as the time from the first documented response (CR or PR) to the earliest relapse or progression
Progression free survival (PFS) | 2 years
  defined as the time from the treatment initiation until the first documented disease progression or death from any cause
Overall survival (OS) | 2 years
  defined as the time from the treatment initiation until death as a result of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Eric Tse, PhD(Cantab), Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong